CLINICAL TRIAL: NCT03736772
Title: A Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3090106 in Japanese and Caucasian Healthy Subjects
Brief Title: A Study of LY3090106 in Japanese and Caucasian Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14828; I6M-JE-SSAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3090106 (Experimental): LY3090106 administered subcutaneously (SC)
  Interventions: Drug: LY3090106
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3090106 — Administered SC
  Arms: LY3090106
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety of a study drug known as LY3090106 in healthy Caucasian and Japanese participants. Side effects and tolerability will be documented. Blood samples will be taken to compare how the body handles the drug. The study will last about 12 weeks, not including screening or additional follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy Japanese or Caucasian
* Body mass index (BMI) 18.0 - 32.0 kilograms per square meter (kg/m²)

Exclusion Criteria:

* Have participated, within the last 30 days, in a clinical study involving an investigational product (IP). If the previous IP has a long half-life, 5 half-lives or 30 days (whichever is longer) should have passed
* Have had symptomatic herpes zoster within 3 months of screening
* Show evidence of active or latent tuberculosis (TB)
* Have known hypogammaglobulinemia or a screening serum immunoglobulin (Ig) G <565 milligrams per deciliter (mg/dL)
* Have received live or attenuated vaccine(s) within 1 month of screening, or intend to during the study
* Are immunocompromised
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing. Participants with any prior exposure to ixekizumab, tabalumab or other biologic agents directly targeting Interleukin 17 (IL-17) and/or B cells (e.g., rituximab, belimumab, etc.) are excluded

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 85
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Maximum Observed Drug Concentration (Cmax) of LY3090106 | Baseline through Day 85
  Cmax of LY3090106
Area Under the Concentration-Versus-Time Curve (AUC) of LY3090106 | Baseline through Day 85
  AUC of LY3090106

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No